CLINICAL TRIAL: NCT05993559
Title: Necessity of Post-mastectomy Radiotherapy in Breast Cancer Patients With an Excellent Response After Neoadjuvant Chemotherapy: A Phase 3, Multicenter, Randomized Controlled Study
Brief Title: Necessity of Post-mastectomy Radiotherapy After Neoadjuvant Chemotherapy and Mastectomy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2023-0178
Record Dates: First submitted 2023-07-20; First posted 2023-08-15 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No PMRT (Experimental): No radiation therapy after neoadjuvant chemotherapy and surgery.
  Interventions: Radiation: Arm I (No PMRT)
- PMRT (Placebo Comparator): Arm Description: Proceed with postoperative radiotherapy, following the guidelines of the respective institution, but advising patients to apply the following points whenever possible.
  * If radiation therapy is administered, include the chest wall and regional LNs.
  * If PMRT field to regional LN, include Axillary LN level III, level IV, Internal mammary LN (1-3rd ICS).
  Interventions: Radiation: Arm II (PMRT)

INTERVENTIONS:
Radiation: Arm I (No PMRT) — The purpose of this study is to confirm that in patients with breast cancer who have undergone mastectomy after prior neoadjuvant chemotherapy, omitting radiotherapy is non-inferior to post-mastectomy radiotherapy (PMRT) in terms of 5-year disease-free survival (DFS) in patients with pathologic complete remission and a good response to treatment corresponding to RCB class 0-I, compared to patients treated with PMRT.
  Arms: No PMRT
Radiation: Arm II (PMRT) — The purpose of this study is to confirm that in patients with breast cancer who have undergone mastectomy after prior neoadjuvant chemotherapy, omitting radiotherapy is non-inferior to post-mastectomy radiotherapy (PMRT) in terms of 5-year disease-free survival (DFS) in patients with pathologic complete remission and a good response to treatment corresponding to RCB class 0-I, compared to patients treated with PMRT.
  Arms: PMRT

SUMMARY:
Postoperative radiotherapy is generally recommended for patients with breast cancer who have undergone breast-conserving surgery, regardless of prior chemotherapy. However, the criteria for postoperative radiation therapy (PMRT) in patients with breast cancer who have received upfront chemotherapy and mastectomy remain controversial. PMRT is recommended for patients with suspected axillary lymph node metastases before chemotherapy or residual cancer in the axillary lymph nodes after surgery, but this varies by institution and physician. In particular, breast cancer patients with a very good treatment response (pCR or RCB 0-I after prior chemotherapy) have a very good prognosis, and the question of whether PMRT is necessary for these patients continues to be raised. With the addition of new targeted therapies and immuno-oncology agents to conventional chemotherapy, the number of patients with good response is increasing, but there are no prospective studies to date.

The studies that have evaluated the need for PMRT in breast cancer patients with a very good treatment response after upfront chemotherapy and mastectomy are all retrospective studies, lacking evidence to apply to standard of care, and have different definitions of a good treatment response group. Therefore, in this study, the investigators aim to reduce unnecessary overtreatment by comparing survival between PMRT and no PMRT in breast cancer patients with a good response to prior chemotherapy and mastectomy, demonstrating non-inferiority of PMRT to no PMRT. By doing so, the investigators hope to reduce patients' side effects and discomfort, improve their satisfaction and quality of life, and contribute to a new standard of care.

The purpose of this study is to confirm that in patients with breast cancer who have undergone mastectomy after prior neoadjuvant chemotherapy, omitting radiotherapy is non-inferior to post-mastectomy radiotherapy (PMRT) in terms of 5-year disease-free survival (DFS) in patients with pathologic complete remission and a good response to treatment corresponding to RCB class 0-I, compared to patients treated with PMRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 20 years of age or older with histologically confirmed invasive breast cancer.
2. Patients with clinical stage IIB-III at the time of diagnosis (including cases of cT1N1 with multiple masses observed during clinical stage IIA). Patients are considered node positive if they have either suspected lymph node metastasis on imaging studies (U/S, breast MRI, PET-CT) or confirmed by pathology.
3. Patients who have undergone mastectomy after prior neoadjuvant chemotherapy.
4. Patients with pathologic complete response (pCR) or residual cancer burden (RCB) class 0-I based on postoperative pathology.

   Complete remission is defined as ypT0/is ypN0. RCB class 0 means complete remission and RCB class 1 is defined as an RCB score ≥0-1.36 as determined by the pathology department at the site.
5. Patients not previously treated for invasive breast cancer.
6. Patients with a systemic performance status of 0-2 based on ECOG.
7. Patients who signed the informed consent prior to study entry.

Exclusion Criteria:

1. Patients with a prior history of invasive breast cancer (patients with a prior history of intraepithelial carcinoma of the breast may be enrolled)
2. Patients with bilateral breast cancer
3. Patients with a prior diagnosis of cancer other than breast cancer within 5 years (however, adequately treated skin cancer other than melanoma and thyroid cancer are eligible for enrollment.)
4. Patients with pathologically or imaging confirmed systemic metastases
5. Patients with a history of prior irradiation or isotope therapy to the rib cage and axillary region contralateral to the breast cancer lesion
6. Patients with suspected supraclavicular/infraclavicular lymph node metastases and internal mammary lymph node metastases
7. Pregnant or lactating patients
8. Patients who have difficulty understanding the contents of the consent form and completing the survey.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2031-04-10 (Estimated); Study Completion 2031-07-10 (Estimated)

PRIMARY OUTCOMES:
5 year invasive disease free survival (iDFS) | 5 year
  Invasive disease-free survival is defined as first invasive recurrence (local, regional, or distant), second invasive cancer (contralateral breast or other cancer), or death from any cause from the date of enrollment.

SECONDARY OUTCOMES:
Overall survival | 5 year
  5-year overall survival (OS): Overall survival is defined as the time from subject enrollment to death from any cause.
Locoregional recurrense free survival | 5 year
  5-year locoregional recurrence-free interval (LRFI): LRFI is defined as the time of first local recurrence of invasive breast cancer from date of enrollment.
Distant metastasis free surviva | 5 year
  5-year distant metastasis-free survival (DMFS): Distant metastasis-free survival is defined as the time from enrollment to the i) first distant metastasis of breast cancer confirmed by imaging (biopsy is performed at the discretion of the investigator). ii) death from breast cancer. iii) death from unknown or non-breast cancer causes.
Complications of radiotherapy | 5 year
  Information on radiotherapy complications including but not restricted to the following items will be collected and any examinations can be ordered at the discretion of the investigator if a patient presents symptoms:
  * Neutropenia
  * Cardiac disease: pericarditis, sinus tachycardia, angina, pericardial effusion, tamponade, cardiac enlargement, heart failure etc.
  * Pulmonary disease: dry cough, dyspnea, pneumonitis etc.
  * Lymphedema of the arm
  * Skin symptoms: erythema, edema, ulceration, hemorrhage, necrosis etc.
  * Esophageal disease: dysphagia, odynophagia, obstruction, ulceration, perforation, fistula etc.